CLINICAL TRIAL: NCT00002598
Title: A PHASE II STUDY OF MITOXANTRONE AND HIGH-DOSE ARA-C FOLLOWED BY INTENSIVE CONSOLIDATION WITH CYCLOPHOSPHAMIDE AND ETOPOSIDE FOR MYELOID BLAST CRISIS OF CHRONIC MYELOGENOUS LEUKEMIA (CML)
Brief Title: Combination Chemotherapy and Interferon Alfa in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 94-070; CDR0000063832 (Registry Identifier: PDQ (Physician Data Query)); NCI-V94-0541
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Blast Crisis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Interferon-alpha; sargramostim; Cyclophosphamide; Cytarabine; Etoposide; Methotrexate; Mitoxantrone; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Procedure: bone marrow ablation with stem cell support
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and interferon alfa in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of induction with high-dose mitoxantrone and cytarabine in patients with chronic myelogenous leukemia (CML) in blast crisis.
* Determine the toxicity and activity of consolidation with high-dose cyclophosphamide and etoposide in these patients.
* Determine the toxicity and activity of maintenance with interferon alfa in these patients.
* Determine the efficacy and tolerability of this regimen in these patients.
* Assess minimal residual disease by cytogenetics, DNA gene rearrangement (Southern blotting), and polymerase chain reaction (PCR) in patients treated with this regimen, and use semiquantitative PCR to evaluate the antileukemic activity of subsequent phases of treatment in patients achieving complete remission.

OUTLINE: Patients are stratified by prior therapy for blast crisis (yes vs no).

* Induction: Patients receive high-dose cytarabine IV over 3 hours on days 1-5 and mitoxantrone IV on day 3. Sargramostim (GM-CSF) is administered subcutaneously (SC) (or IV over 4 hours) daily beginning on day 7 and continuing until blood counts recover. After completion of induction, patients with a suitable HLA-identical bone marrow donor undergo allogeneic bone marrow transplantation according to an appropriate IRB-approved protocol. Patients without a donor proceed to consolidation approximately 4 weeks after hospital discharge following induction.
* Consolidation: Patients receive high-dose cyclophosphamide IV on days 1-4 and etoposide IV continuously on days 5-7. GM-CSF is administered SC (or IV over 4 hours) beginning on day 8 and continuing until blood counts recover. Patients achieving a second chronic phase or complete remission proceed to maintenance approximately 4 weeks after hospital discharge following consolidation.
* Maintenance: Patients receive interferon alfa SC on day 1. Treatment with interferon alfa continues daily in the absence of disease progression or unacceptable toxicity.

Patients with CNS involvement at entry or who develop CNS disease during the study receive CNS therapy as outlined below.

* CNS therapy: Patients undergo whole brain irradiation as soon as possible but not concurrently with mitoxantrone. Patients also receive methotrexate intrathecally 3 times a week until the CSF is clear, weekly for 4 weeks, and then monthly for 6 months.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia in blast crisis

  * Bone marrow blasts at least 20% OR
  * Bone marrow blasts plus promyelocytes at least 50%
* Ineligible for higher priority protocols

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* LVEF greater than 50% by MUGA scan or echocardiogram

Other:

* HIV negative
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Prior therapy for blast crisis allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1994-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Adam Weiss, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States